CLINICAL TRIAL: NCT06986863
Title: Use of a Digital Snapshot to Reduce Use of Restraints During Emergency Department Visits and Improve Experience of Care for PWIDD
Acronym: SCANS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Institute for Exceptional Care (Unknown)
Responsible Party: Principal Investigator, Sophia Jan, Division Chief, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-0125
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Intellectual and Developmental Disabilities
Keywords: Intellectual and developmental disabilities; emergency department; restraint; restraint, physical; emergency department visits
MeSH Terms: conditions — Developmental Disabilities; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): This arm will not be given any interventions.
- Always Uniquely Me (AUM) arm (Experimental): Participants will receive access to the Always Uniquely Me app.
  Interventions: Other: Always Uniquely Me mobile phone application

INTERVENTIONS:
Other: Always Uniquely Me mobile phone application — The app will allow the user to organize their healthcare information and personal needs which can help improve communication with doctors, clinicians and first responders.
  Arms: Always Uniquely Me (AUM) arm

SUMMARY:
The purpose of this research study is to compare the Always Uniquely Me (AUM) mobile application to regular medical care. The investigators want to know if AUM is helpful at decreasing use of restraints and improving experience in the emergency department (ED) for people with intellectual and developmental disabilities (PWIDD). The investigators will also be looking at how certain characteristics of the PWIDD participants may affect those outcomes.

DETAILED DESCRIPTION:
PWIDD have high rates of ED use and poor quality of experience in EDs compared to the general population. Among a multistate cohort of adults with IDD, the risk of emergency department visits for adults with IDD was more than twice that for other adults, particularly for conditions that can be safely treated in the community (e.g., urinary tract and respiratory infections), and psychiatric conditions.1 PWIDD were more likely than those without IDD to visit the ED in a population based cohort in Ontario, Canada. For both groups, receiving greater continuity of primary care was associated with less ED use, but this relationship was more marked for adults with IDD. Another national study also found that compared to children with IDD with no emergency room visits, those with 3 or more emergency room visits were less likely to report access to a source of outpatient healthcare.

PWIDD have poor experiences in EDs. A large survey of PWIDD recently admitted to a hospital who were recruited from disability service organizations found that 12% did not always get the right medication; 22% didn't get their medication on time or only sometimes; 18% didn't get enough to drink; 13% didn't get enough to eat; 39% could not get to the toilet when they needed to, while 7% could do so only sometimes; and 11% reported not getting help in moving from their bed when needed. A systematic review of hospital experiences of people with intellectual disability found similar findings, citing failures of hospitals and staff to meet patient needs due to limited knowledge and skills of staff, negative attitudes, hospital systems failing to make required adjustments, and reliance on carers for both care and advocacy for appropriate treatment.

There is some evidence that tools like AUM improve PWIDD's experiences and outcomes.

Patient-held medication lists may improve experience by (a) creating the "glue" between disjointed healthcare systems, (b) enhancing situational awareness among clinical teams, (c) support clinical teams in checking for errors, (d) ease challenges in communication, (e) improve patient empowerment, (f) serve as a memory aide during appointments when patients are under stress, (g) serve as a reminder to take medications, and (h) serve as a reminder for clinicians to reorder medications.

Among people with diabetes undergoing surgery, those randomized to use of health passports similar to AUM received more information about their expected diabetes care prior to surgery (92% vs 35%), were more involved in planning their diabetes care, were less anxious while in the hospital, more prepared to manage their diabetes care on discharge, and had a shorter mean length of stay (4.4 vs 6.5 days) compared to controls. Among people with diabetes in New Zealand, use of a health passport was associated with a relative reduction in HbA1c of 0.4% (a measure of diabetes control) and a relative increase in weight of 1.0 kg/m2, but no changes in diabetes knowledge, attitudes to diabetes or risk factors for diabetic tissue damage. In another study of adults with diabetes followed in nine Dutch general hospitals, use of a healthcare passport let to small but significant changes in mean HbA1c levels.

There is no published evidence on the impact of health passports on use of restraints during ED visits in any population. Among individuals with congenital heart disease, a health passport showed initial improvements in disease knowledge or physical activity intensity, but those effects were not sustained at 6 months or 1 year. Among individuals with inflammatory bowel disease, health passports and Standardized routine email interactions between an IBD nurse and patients does not reliably improve most traditional disease outcomes. Among individuals with rheumatoid arthritis, there were no effects on self-efficacy expectations, knowledge, health status, or behavior among those with and without health passports.

Because previous studies have shown mixed results of using health passports and other tools similar to AUM, and no prior studies have examined their impact in particular on the use of restraints during ED visits, it is important to systematically collect new data for analysis to determine whether this tool will meaningfully reduce rates of use of restraints during ED visits, and improve the experience of PWIDD, their care partners.

Compelling data and rigorous evaluation findings will allow clinics, hospitals and health systems, insurers, disability service organizations, and public agencies like Medicaid or departments for developmental disabilities to make informed decisions about whether/how to expand use of the tool. Findings from this evaluation will also support stakeholders in developing business cases for covering use of the tool as a benefit, whether in an insurance product or as part of government or community programs.

The investigators will conduct a two-arm, pragmatic randomized controlled trial (RCT) of PWIDD, who will be randomized 1:1 to either to standard care plus AUM, or to the control group that will receive standard care and will not have access to the tool stratified by PWIDD or proxy respondent status and presence of maladaptive behaviors. This is a non-blinded study because the nature of the intervention prevents participants from being blinded to their study arm. The primary goal of this study is to compare the effectiveness of the AUM mobile app vs. standard care on the use of restraints and experience of PWIDD and their care partners in the ED and in other clinical settings.

The study team will recruit potential participants who have engaged with any Northwell Health emergency department in the previous 12 months. The team's goal is to enroll 1,500 eligible PWIDD. If participants are unable to answer questions on their own, legally authorized representative will be engaged to provide proxy responses. Primary research participants will be asked to identify an individual who assists with medical care (care partner). Care partners will be approached for participation as secondary research subjects and will answer survey questions about their own experience while caring for their PWIDD care recipient in ED and ambulatory settings.

ELIGIBILITY:
Inclusion criteria for primary participant/PWIDD (person with intellectual and/or developmental disability):

* have visited a Northwell Health Emergency Department in the last 12 months
* have a confirmed intellectual and/or developmental disability
* must be 18 years of age or older at enrollment
* have a smart phone or tablet that connects to the internet
* have a preferred language of English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Use of physical and/or chemical restraints during ED visits | 12 months
  Measured using electronic medical record data.

SECONDARY OUTCOMES:
Length of stay in the ED | 12 months
  Captured using electronic medical record data.
Experience of care in hospital-based EDs | Baseline, 6 months, 12 months
  Measured through the Emergency Department Consumer Assessment of Healthcare Providers and Systems (ED CAHPS). The questions were modified for reading level of the respondent and appropriateness for the study. This includes 17-19 questions that require yes/no, Likert Scale, and select-all-that-apply answers.

OTHER OUTCOMES:
Perceptions of self and publicly enacted negativity, prejudice, and discrimination | Baseline, 6 months, 12 months
  Measured through the Quality of Life In Neurological Disorders Measurement System - stigma short form (Neuro-QoL stigma SF), a validated survey that includes 8 questions with Likert scale answer choices.
Perceived functional communication abilities | Baseline, 6 months, 12 months
  Measured through Quality of Life In Neurological Disorders Measurement System - communication short form (Neuro-QoL communication SF), a validated survey that includes 5 questions with Likert scale answer choices.
Overall health status, including physical, mental, and social health | Baseline, 6 months, 12 months
  Measured through the Patient-Reported Outcomes Measurement Information Systems Global Health (PROMIS global health), a validated survey that includes 10 questions with Likert scale answer choices.
Perceived usability of the mobile health application | Baseline, 6 months, 12 months
  Measured by the System Usability Scale (SUS). This is a validated survey with 10 questions that use Likert Scale answer choices. On yes/no question was added to capture perceived usage of the mobile app.
Experience of care in urgent care settings, including virtual visits | Baseline, 6 months, 12 months
  Measured through the Clinician and Group Consumer Assessment of Healthcare Providers and Systems (CG CAHPS). The questions were modified to address experiences in the urgent care setting, for reading level of respondent, and appropriateness for the study. This includes 20-22 questions that require yes/no, Likert Scale, and select-all-that-apply answers.
Experience of care in outpatient doctor and clinic settings, including virtual visits | Baseline, 6 months, 12 months
  Measured through the Clinician and Group Consumer Assessment of Healthcare Providers and Systems (CG CAHPS). The questions were modified to address experiences in the outpatient clinic, for reading level of respondent, and appropriateness for the study. This includes 20-22 questions that require yes/no, Likert Scale, and select-all-that-apply answers.
Confidence in managing daily activities | Baseline, 6 months, 12 months
  Measured through the Patient-Reported Outcomes Measurement Information Systems Self Efficacy (PROMIS self-efficacy), a validated survey that includes 8 questions with Likert scale answer choices.
Perceived functional impairments during wakefulness associated with sleep problems | Baseline, 6 months, 12 months
  Measured by the Patient-Reported Outcomes Measurement Information Systems - Sleep-Related Impairment (PROMIS Short Form v1.0 - Sleep-Related Impairment - Short Form 4a), a validated survey that includes 4 questions with Likert Scale answer choices.
Perceived sleep quality, depth, and restoration | Baseline, 6 months, 12 months
  Measured by the Quality of Life In Neurological Disorders Measurement System - Sleep Disturbance (Neuro-QOL Item Bank v1.0 - Sleep Disturbance - Short Form), a validated survey that includes 8 questions with Likert Scale answer choices.
Symptoms associated with stomach contents leaking backwards from the stomach into the esophagus | Baseline, 6 months, 12 months
  Measured by the Patient-Reported Outcomes Measurement Information Systems - Gastrointestinal Gastroesophageal Reflux (PROMIS® Scale v1.0 - Gastrointestinal Gastroesophageal Reflux 13a), a validated survey that includes 13 questions with Likert Scale answer choices.
Frequency and intensity of incomplete evacuation, rectal pain, straining, and hard stools | Baseline, 6 months, 12 months
  Measured by the Patient-Reported Outcomes Measurement Information Systems - Gastrointestinal Constipation (PROMIS Scale v1.0 - Gastrointestinal Constipation 9a), a validated survey that includes 9 questions with Likert Scale answer choices.
Impact of emotional and behavioral difficulties on the health-related quality of life | Baseline, 6 months, 12 months
  Measured by the Quality of Life In Neurological Disorders Measurement System- Emotional and Behavioral Dyscontrol (Neuro-QOL Item Bank v1.0 - Emotional and Behavioral Dyscontrol - Short Form), a validated survey that includes 8 questions with Likert Scale answer choices.
Negative mood, views of self, and social cognition, as well as decreased positive affect and engagement | Baseline, 6 months, 12 months
  Measured by the Patient-Reported Outcomes Measurement Information Systems - Depression (PROMIS® Item Bank v1.0 - Emotional Distress-Depression - Short Form 4a), a validated survey that includes 4 questions with Likert Scale answer choices.
Fear, anxious misery, hyperarousal , and somatic symptoms related to arousal | Baseline, 6 months, 12 months
  Measured by the Patient-Reported Outcomes Measurement Information Systems - Emotional Distress-Anxiety (PROMIS Item Bank v1.0-Emotional Distress-Anxiety - Short Form 4a), a validated survey that includes 4 questions with Likert Scale answer choices.

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riemsma RP, Taal E, Brus HL, Rasker JJ, Wiegman O. Coordinated individual education with an arthritis passport for patients with rheumatoid arthritis. Arthritis Care Res. 1997 Aug;10(4):238-49. doi: 10.1002/art.1790100405. PMID 9295453
- [Background] Lin PJ, Fanjiang YY, Wang JK, Lu CW, Lin KC, Cheong IM, Pan KY, Chen CW. Long-term effectiveness of an mHealth-tailored physical activity intervention in youth with congenital heart disease: A randomized controlled trial. J Adv Nurs. 2021 Aug;77(8):3494-3506. doi: 10.1111/jan.14924. Epub 2021 Jun 21. PMID 34151444
- [Background] Valente AM, Landzberg MJ, Gianola A, Harmon AJ, Cook S, Ting JG, Stout K, Kuehl K, Khairy P, Kay JD, Earing M, Houser L, Broberg C, Milliren C, Opotowsky AR, Webb G, Verstappen A, Gurvitz M; Alliance for Adult Research in Congenital Cardiology (AARCC) Investigators; Adult Congenital Heart Association (ACHA). Improving heart disease knowledge and research participation in adults with congenital heart disease (the Health, Education and Access Research Trial: HEART-ACHD). Int J Cardiol. 2013 Oct 9;168(4):3236-40. doi: 10.1016/j.ijcard.2013.04.004. Epub 2013 May 4. PMID 23651823
- [Background] Murphy P, Levine A, Lerma T, Young S, Hwang J, Goldsby R. A portable survivorship care plan: a tool that helps educate and improve knowledge in childhood cancer survivors. Support Care Cancer. 2021 Jan;29(1):169-177. doi: 10.1007/s00520-020-05422-z. Epub 2020 Apr 23. PMID 32328773
- [Background] Simmons D, Gamble GD, Foote S, Cole DR, Coster G; New Zealand Diabetes Passport Study. The New Zealand Diabetes Passport Study: a randomized controlled trial of the impact of a diabetes passport on risk factors for diabetes-related complications. Diabet Med. 2004 Mar;21(3):214-7. doi: 10.1111/j.1464-5491.2004.01047.x. PMID 15008829
- [Background] Page E, Akiboye F, Jackson S, Kerry C, Round R, Rayman G; DICE team*. Perioperative passport: empowering people with diabetes along their surgical journey. Diabet Med. 2017 Dec;34(12):1737-1741. doi: 10.1111/dme.13513. Epub 2017 Oct 20. PMID 28921676
- [Background] Garfield S, Furniss D, Husson F, Etkind M, Williams M, Norton J, Ogunleye D, Jubraj B, Lakhdari H, Franklin BD. How can patient-held lists of medication enhance patient safety? A mixed-methods study with a focus on user experience. BMJ Qual Saf. 2020 Sep;29(9):764-773. doi: 10.1136/bmjqs-2019-010194. Epub 2020 Jan 16. PMID 31949006
- [Background] Iacono T, Bigby C, Unsworth C, Douglas J, Fitzpatrick P. A systematic review of hospital experiences of people with intellectual disability. BMC Health Serv Res. 2014 Oct 25;14:505. doi: 10.1186/s12913-014-0505-5. PMID 25344333
- [Background] Iacono T, Davis R. The experiences of people with developmental disability in Emergency Departments and hospital wards. Res Dev Disabil. 2003 Jul-Aug;24(4):247-64. doi: 10.1016/s0891-4222(03)00041-6. PMID 12873658
- [Background] Lin SC, Margolis B, Yu SM, Adirim TA. The role of medical home in emergency department use for children with developmental disabilities in the United States. Pediatr Emerg Care. 2014 Aug;30(8):534-9. doi: 10.1097/PEC.0000000000000184. PMID 25062298
- [Background] Durbin A, Balogh R, Lin E, Wilton AS, Lunsky Y. Emergency Department Use: Common Presenting Issues and Continuity of Care for Individuals With and Without Intellectual and Developmental Disabilities. J Autism Dev Disord. 2018 Oct;48(10):3542-3550. doi: 10.1007/s10803-018-3615-9. PMID 29923146
- [Background] Lauer E, Lindgren S, Momany E, Cope T, Royer J, Cogan L, McDermott S, Armour B. Health Service Utilization Patterns Among Medicaid-Insured Adults With Intellectual and Developmental Disabilities: Implications for Access Needs in Outpatient Community-Based Medical Services. J Ambul Care Manage. 2021 Apr-Jun 01;44(2):138-147. doi: 10.1097/JAC.0000000000000373. PMID 33492884
- See also: Unity Health Toronto. Exploring the Efficacy and Usability of the My Autism Passport (MAP) App in Service Navigation for Families of Children With Autism. clinicaltrials.gov; 2020. Accessed January 16, 2023. — https://clinicaltrials.gov/ct2/show/NCT04259671
- See also: Bollegala N, Lomonaco J, Colucci A, et al. A85 IMPROVING OUTCOMES IN THE PEDIATRIC TO ADULT CARE TRANSITION IN IBD (IMPACT IBD). J Can Assoc Gastroenterol. 2019;2(Supplement_2):169-170. doi:10.1093/jcag/gwz006.084 — https://pmc.ncbi.nlm.nih.gov/articles/PMC6512494/